CLINICAL TRIAL: NCT02599792
Title: A Two-Part Phase 1 Healthy Volunteer Study: A Crossover Comparison of CTP-656 Solid Dose Formulation vs. Kalydeco® and a Double-Blind, Placebo-Controlled, Ascending Multiple Dose Evaluation of CTP-656
Brief Title: Healthy Volunteer Solid Oral Dose and Multiple Ascending Dose Evaluation of CTP-656
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CP656.1002
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: Safety and Pharmacokinetics
MeSH Terms: interventions — ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- CTP-656, 150 mg (Experimental): Single Oral Dose
  Interventions: Drug: CTP-656
- Kalydeco, 150 mg (Active Comparator): Single oral dose
  Interventions: Drug: Kalydeco
- CTP-656, 75 mg or matching placebo (Experimental): Subjects will be administered 75 mg CTP-656 for 7 days.
  Interventions: Drug: CTP-656; Drug: Placebo for CTP-656
- CTP-656, 150 mg or matching placebo (Experimental): Subjects will be administered 150 mg CTP-656 for 7 days.
  Interventions: Drug: CTP-656; Drug: Placebo for CTP-656
- CTP-656, high dose or matching placebo (Experimental): Subjects will be administered up to 300 mg CTP-656 for 7 days.
  Interventions: Drug: CTP-656; Drug: Placebo for CTP-656

INTERVENTIONS:
Drug: CTP-656
  Arms: CTP-656, 150 mg; CTP-656, 150 mg or matching placebo; CTP-656, 75 mg or matching placebo; CTP-656, high dose or matching placebo
Drug: Placebo for CTP-656
  Arms: CTP-656, 150 mg or matching placebo; CTP-656, 75 mg or matching placebo; CTP-656, high dose or matching placebo
Drug: Kalydeco
  Arms: Kalydeco, 150 mg

SUMMARY:
Two-part study to assess CTP-656 dosed as a solid oral dosage form versus Kalydeco and multiple-ascending doses of CTP-656 dosed for 7 days.

DETAILED DESCRIPTION:
This two-part study will assess in healthy male and female subjects a solid oral dose formulation of CTP-656 vs. Kalydeco® and the safety, tolerability and pharmacokinetic profiles of escalating CTP-656 solid oral doses following 7 days of dosing. In Part B, three doses of CTP-656 ranging from 75 mg up to 300 mg per day will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between 18 and 50 years of age, inclusive
* Body weight ≥ 50 kg and BMI within the range of 18 to 30 kg/m2, inclusive, at screening

Exclusion Criteria:

* History of clinically significant central nervous system (eg, seizures), cardiac, pulmonary, metabolic, renal (including nephrolithiasis), hepatic, including history of Gilbert's syndrome or gastrointestinal (GI) conditions
* PR interval ≥ 220 msec or QRS duration ≥ 120 msec or QTcF interval > 450 msec obtained at screening visit or prior to the first dose of study drug
* Liver function tests greater than the upper limit of normal.
* Positive blood screen for human immunodeficiency virus (HIV antibody), hepatitis B virus surface antigen, or hepatitis C virus antibody at screening
* Urinalysis positive for greater than trace blood, protein or glucose
* A positive screen for alcohol, drugs of abuse, or tobacco use.
* Inability to comply with food and beverage restrictions during study participation.
* Donation or blood collection or acute loss of blood prior to screening.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 7 days
  adverse events categorized by body system and MedDRA term
Measure exposure of test articles using area under the concentration time curve (AUC) | 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Lana Pilja, Study Director — Concert Pharmaceuticals, Inc.
Locations (1):
- Adelaide, South Australia, Australia